CLINICAL TRIAL: NCT00250666
Title: Procalcitonin-Guided Antimicrobial Discontinuation Strategy in Critically Ill Patients With Suspected or Confirmed Bacterial Sepsis
Brief Title: Procalcitonin-Guided Antimicrobial Discontinuation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HUG 05-146
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Sepsis
Keywords: Biological Markers; Procalcitonin; Critical Care; Diagnosis, Differential; Prospective Study; Sepsis; Antibiotic stewardship; Antimicrobial resistance
MeSH Terms: conditions — Sepsis; Disease

INTERVENTIONS:
Procedure: PCT measurement — Peripheral blood samples were collected in the morning, using vacuum tubes (BD Vacutainer SST II Plus plastic tubes; Becton Dickinson Diagnostic Systems, Allschwil, Switzerland). Circulating plasma PCT levels were measured with a time-resolved amplified cryptate emission technology assay (Kryptor PCT; Brahms AG, Hennigsdorf, Germany), with an assay sensitivity of 0.06 mg/L, approximately fourfold above mean normal levels. Measurements were performed 7 days a week.

SUMMARY:
The current study aims to validate the diagnostic use of PCT assessing its capability to individualize and shorten the duration of antibiotic therapy in critically ill patients with suspected or confirmed sepsis.

In particular, no well-designed intervention study has properly examined the following hypothesis: A PCT-guided antibiotic discontinuation strategy enables to reduce antibiotic treatment duration in critically ill patients with suspected or documented sepsis, without harming patient safety.

DETAILED DESCRIPTION:
Primary objective:

To assess the effect of repeated PCT measurements in critically ill patients with clinically suspected or microbiologically documented sepsis on duration of antimicrobial use and to compare this strategy to standard clinical practice, by using an improved PCT assay with a sensitivity of 0.06 ng/ml.

Secondary objectives:

To determine the impact of repeated PCT measurements on patient outcome (morbidity, mortality, emergence of antibiotic resistance and nosocomial super-infections).

Main measures:

Primary:

1. Exposure to systemic antimicrobial treatment (in duration of antibiotic treatment and total antibiotic exposure)

   Secondary:
2. Cure and failure rate of infection (in N recurrent infections per 100 patients)
3. 28-day case-fatality rate (in N deaths per 100 patients)
4. Length of hospital stay (in days)
5. Costs of antimicrobial therapy (in CHF)
6. Rate of nosocomial super-infection (in N super-infections per 100 patients)
7. Isolation of multi-resistant microorganisms (in clinical isolates per 100 patient-days)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically suspected or microbiologically confirmed bacterial sepsis
2. Informed consent

Exclusion Criteria:

1. Patients with microbiologically documented infections caused by the following microorganisms: Listeria spp, Legionella pneumophilia, Mycobacterium tuberculosis, Staphylococcus aureus
2. Patients with fungal infections
3. Patients with severe infections due to viruses or parasites (e.g. hemorrhagic fever, malaria)
4. Patients with suspected or confirmed bacterial meningitis or endocarditis
5. Patients with localized, deep-seated abscesses (e.g. brain abscess) without systemic sepsis
6. Patients with chronic, localized infections (e.g. chronic osteomyelitis) without systemic sepsis
7. Neutropenic and other severely immuno-compromised patients (patients infected with human immunodeficiency virus and a CD4 count < 200; patients on immuno-suppressive therapy after solid organ transplantation; patients with cystic fibrosis)
8. Withholding of life-support
9. Early discharge or death (< 24 hours after admission)
10. Complete absence of antimicrobial treatment despite suspicion of sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Exposure to systemic antimicrobial treatment (in duration of antibiotic treatment and total antibiotic exposure)

SECONDARY OUTCOMES:
Cure and failure rate of infection (in N recurrent infections per 100 patients)
28-day case-fatality rate (in N deaths per 100 patients)
Length of hospital stay (in days)
Costs of antimicrobial therapy (in CHF)
Rate of nosocomial super-infection (in N super-infections per 100 patients)
Isolation of multi-resistant microorganisms (in clinical isolates per 100 patient-days)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan J Harbarth, MD MS, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva Universits Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708